CLINICAL TRIAL: NCT02174237
Title: LNP1892 - A Phase I, Double-Blind, Placebo-Controlled, Ascending Single and Multiple Oral Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Healthy Male and Female Subjects
Brief Title: A Study to Test the Safety/Tolerability of Increasing Doses of LNP1892 Versus Placebo in Healthy Male/Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRP/LNP1892/2014/001; 2014-000327-24 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Phase 1, safety, tolerability, PK, PD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LNP1892 (Experimental): Dosage Form: Tablet Two Parts. Part A: Single Ascending Dose (SAD) starting with 25 mg (Maximum 5 cohorts). Part B: Multiple Ascending Dose (MAD), 10 days dosing, Maximum 3 cohorts. Six subjects in each cohort will receive LNP1892
  Interventions: Drug: LNP1892
- Placebo (Placebo Comparator): Two subjects in each cohort will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LNP1892 — Tablets of two strengths (5 and 25 mg)
  Arms: LNP1892
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple ascending oral dose LNP1892 in healthy males and female subjects

DETAILED DESCRIPTION:
This is first in human, Phase 1 study. Primary purpose is to assess safety, tolerability, pharmacodynamic and pharmacokinetic of the LNP1892. Study will be conducted in healthy human subjects. Pharmacokinetic will be studied in the subjects after administration of single and multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be; males or females (Group A3 only), of any ethnic origin, between 18 and 65 years of age (both inclusive)
* Subjects will have a body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive
* Subjects must be in good health, as determined by; medical history, physical examination, vital sign assessment, 12-lead electrocardiogram (ECG)
* Clinical laboratory evaluations (congenital non-haemolytic hyperbilirubinaemia is not acceptable)
* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

* Male subjects who are not willing, or whose partners are not willing, to use appropriate contraception until 3 months after the final dosing occasion.
* Female subjects who are of child-bearing potential; or those with tubal ligation.
* Subjects who have donated; blood in the 3 months prior to screening, plasma in the 7 days prior to screening, platelets in the 6 weeks prior to screening
* Subjects who;consume alcohol, cigarettes, tobacco and have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator
* Subjects who have used any non-prescribed systemic or topical medication, herbal remedies, Vitamin supplements, mineral supplements within 7 days of the first dose administration.
* Subjects who have received any medications, within 30 days of the first dose administration, or any prescribed systemic or topical medication within 14 days of the first dose administration
* Subjects who have an abnormality in heart rate, blood pressure, temperature or respiration rate.
* Subjects with; a positive urine drug screen, a positive alcohol breath test result at screening or first admission.
* Subjects who have an abnormality in the 12-lead ECG.
* Female subjects who are pregnant or lactating
* Subjects who are participating in a clinical study or who have participated in a clinical study involving administration of an investigational drug (new molecular entity) in the past 3 months.
* Subjects with a significant history of drug allergy to similar drug or its excipients.
* Subjects who have any clinically significant medical history or significant allergic condition in the opinion of the investigator
* Subjects with clinically significant out of range PTH or serum calcium or vitamin D levels as judged by the investigator. Subjects with current or a history of hypocalcaemia
* Subjects who; are known to have serum hepatitis, are carriers of the hepatitis B surface antigen (HBsAg) are carriers of the hepatitis C antibody, have a positive result to the test for HIV antibodies.
* Subjects who have previously taken part in or withdrawn from this study post first drug administration.
* Other standard exclusion criteria like Subjects who have a clinically significant disorder or a significant abnormal laboratory finding, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of single and multiple oral doses of LNP1892 in healthy subjects | Up to 30 days after last dose

SECONDARY OUTCOMES:
To determine the single and multiple oral dose pharmacokinetics of LNP1892 in healthy subjects | Pre-dose to 72 hours post last dose
To determine the single and multiple oral dose pharmacodynamics of LNP1892 in healthy subjects. | Pre-dose to 72 hours post last dose

OTHER OUTCOMES:
Exploratory Objectives: To determine the effect of food on the single oral dose pharmacokinetics of LNP1892 in healthy subjects | Pre-dose to 72 hours post last dose
Exploratory Objectives: To determine the effect of gender on the single oral dose pharmacokinetics of LNP1892 in healthy subjects | Pre-dose to 72 hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MB ChB, PhD, Study Director — Covance
Locations (1):
- Covance Clinical Research Unit Ltd. Springfield House Hyde Street, Leeds, United Kingdom